CLINICAL TRIAL: NCT01700348
Title: An Investigation of the Effects of a Oral Hygiene Regimen in Irregular Flossers on Gingivitis and Plaque
Brief Title: Philips AirFlosser Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated by financier due to low accrual & high number of protocol deviations.
Sponsor: Tufts University (Other)
Collaborators: Philips Oral Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAH-12-0081; 10438 (Other: TUSDM IRB)
Record Dates: First submitted 2012-08-20; First posted 2012-10-04 (Estimated); Results first posted 2015-05-29 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Gingivitis
Keywords: moderate gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Airflosser (Experimental): Use of Airflosser
  Interventions: Device: Airflosser
- Manual Floss (Active Comparator): Normal Routine
  Interventions: Device: Manual Floss

INTERVENTIONS:
Device: Airflosser — Use of Philips Airflosser
  Other Names: Philips Airflosser
  Arms: Airflosser
Device: Manual Floss — Active Comparator
  Arms: Manual Floss

SUMMARY:
In the current study, Sonicare AirFloss (AF) will be used in combination with a Manual Toothbrush (MTB) in a population of manual toothbrush users who are irregular flossers and who exhibit signs of moderate gingivitis. The alternate test arm will be allocated to a No Intervention group and will be given no test products or instruction other than to change none of their typical at home oral hygiene habits.

The aim of this study is to investigate how an AF and MTB oral hygiene intervention will affect a population of irregular flossers using the residual protein concentration method as an interproximal plaque efficacy assessment. Gingivitis reduction will be assessed using the Modified Gingival Index (MGI) and Gingival Bleeding Index (GBI) indices

ELIGIBILITY:
4.1 Inclusion Criteria

Subjects accepted into the study must meet the following requirements:

* are 18-70 years;
* are in generally good health;
* have a minimum of 20 natural teeth (excluding 3rd molars);
* have 1 qualifying test site in each posterior quadrant;
* are a regular manual toothbrush user (prior periodic use of powered toothbrushes in other studies permitted);
* Irregular Flossers defined as using dental floss ≤ 2 days a week;
* be willing and able to comply with study procedures and be available at all times required for participation;
* have a Gingival Bleeding Index > 1 on at least 20 sites;
* be a non-smoker.

4.2 Exclusion Criteria Subjects will be excluded from the study if they;

* have systemic diseases such as Down's syndrome, or known AIDS/HIV;
* have insulin dependent Diabetes;
* are pregnant or nursing by subject report;
* have a cardiac pacemaker or AICD;
* are undergoing or require extensive dental or orthodontic treatment;
* require antibiotic treatment for dental appointments;
* have used antibiotics within 4 weeks of enrollment;
* are currently using prescription-dose anti-inflammatory medications or anticoagulants (including aspirin);
* have heavy deposits of calculus, either supragingival and/or subgingival;
* have severe gingivitis or periodontitis;
* have extensive crown or bridge work and/or rampant decay;
* are currently use bleaching trays;
* have any oral or extraoral piercing on lips or in mouth with ornament or accessory;
* have a professional prophylaxis within 4 weeks of study;
* have participated in a prior study ≤ 20 days;
* are employed by an oral healthcare products company or dental research institution.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2012-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Kugel, DMD, MS, PhD, Principal Investigator — TUSDM
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 257 subjects who signed consent forms, 140 (54.5% were classified as screen failures). 1 additional subject declined to participate after screening but before randomization.
Groups:
- All Enrolled Subjects: Airflosser & Manual Floss
Period: Overall Study
Arm/Group | All Enrolled Subjects
Started | 116
Completed | 93
Not Completed | 23
Not completed — Withdrawal by Subject | 22
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Data cannot be provided for each arm separately, but only in aggregate
Groups:
- All Randomized Subjects: The study was terminated early, data were not analyzed and the plaque samples were destroyed. Data cannot be provided for each arm separately, but only in aggregate.
Arm/Group | All Randomized Subjects
Number analyzed (Participants) | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 116
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (11.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 42
Region of Enrollment [Number; unit: participants]
  United States | 116
Number of Missing Teeth [Mean (Standard Deviation); unit: missing teeth] | .8 (1.40)
Average Modified Gingival Index Score [Mean (Standard Deviation); unit: units on a scale] — The Modified Gingival Index (MGI) scale 0 = absence of inflammation;
  1. = mild inflammation or with slight changes in color and texture but not in all portions of gingival marginal or papillary;
  2. = mild inflammation, such as the preceding criteria, in all portions of gingival marginal or papillary;
  3. = moderate, bright surface inflammation, erythema, edema and/or hypertrophy of gingival marginal or papillary;
  4. = severe inflammation: erythema, edema and/or marginal gingival hypertrophy of the unit or spontaneous bleeding, papillary, congestion or ulceration.
  units on a scale | 1.2 (.4)
Number of Bleeding Sites [Mean (Standard Deviation); unit: number of sites] | 54.1 (17.80)
Percent of Site Bleeding [Mean (Standard Deviation); unit: percent of sites] | 51.6 (16.70)

OUTCOME MEASURES:

1. Primary Outcome: The Effect of Sonicare AirFloss + MTB Treatment Versus the Control Group
Description: The primary objective of the study is to compare the effect of Sonicare AirFloss + MTB treatment versus the Control Group on gingival inflammation (as measure by number of bleeding sites, and reduction in MGI) after four weeks of use.
Time Frame: Four Months
Population: Terminated by financier due to low accrual & high number of protocol deviations.
Groups:
- All Randomized Subjects: The study was terminated early, data were not analyzed and the plaque samples were destroyed."
Arm/Group | All Randomized Subjects
Number analyzed (Participants) | 0

2. Secondary Outcome: Gingival Inflammation
Description: Evaluate the effect of the Sonicare AirFloss + MTB treatment on gingival inflammation as measured after 2 and 4 weeks versus baseline.
Time Frame: 4 weeks
Population: The study was terminated early, data were not analyzed and the plaque samples were destroyed.
Groups:
- All Randomized Subjects: The study was terminated early, data were not analyzed and the plaque samples were destroyed.
Arm/Group | All Randomized Subjects
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Bleeding Sites
Description: Compare the number of bleeding sites in Modified Gingival Index following 2 weeks of use of the Sonicare AirFloss + Manual Toothbrush versus the Control Group.
Time Frame: 2 Weeks
Population: The study was terminated early, data were not analyzed and the plaque samples were destroyed.
Arm/Group | All Randomized Subjects
Number analyzed (Participants) | 0

4. Secondary Outcome: Plaque
Description: Compare plaque as measured by the reduction and percent reduction in Residual Protein Concentration (RPC) following 2 and 4 weeks of use of the Sonicare AirFloss + MTB and Control Group.
Time Frame: 4 Weeks
Population: The study was terminated early, data were not analyzed and the plaque samples were destroyed.
Arm/Group | All Randomized Subjects
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Assess the safety of the Sonicare AirFloss + MTB treatment.
Time Frame: 4 Months
Population: The study was terminated early, data were not analyzed and the plaque samples were destroyed.
Arm/Group | All Randomized Subjects
Number analyzed (Participants) | 0

6. Secondary Outcome: Percentage of Bleeding Sites
Description: Compare the percentage of bleeding sites in Modified Gingival Index following 2 weeks of use of the Sonicare AirFloss + Manual Toothbrush versus the Control Group.
Time Frame: 2 Weeks
Population: The study was terminated early, data were not analyzed and the plaque samples were destroyed.
Arm/Group | All Randomized Subjects
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- All Randomized Subjects: Summary of AEs for All Randomized Subjects
Arm/Group | All Randomized Subjects
Serious Adverse Events (participants affected / at risk) | 0/116
Other Adverse Events (participants affected / at risk) | 0/116

LIMITATIONS AND CAVEATS:
Terminated by sponsor due to:

* Changes in business strategy/Target completion dates not being met
* Higher than anticipated screen failure rate
* Higher than anticipated early termination rate
* Large number of protocol deviations encountered

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less